CLINICAL TRIAL: NCT04553211
Title: Expedited Partner Therapy and the HIV Prevention Cascade for MSM in Peru
Brief Title: Expedited Partner Therapy and the HIV Prevention Cascade
Acronym: EPT and MSM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Asociación Civil Via Libre, Peru (Other); University of California, San Francisco (Other); Emory University (Other)
Responsible Party: Principal Investigator, Jesse Clark, Associate Professor-in-Residence, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01MH118973 (NIH)
Record Dates: First submitted 2020-09-06; First posted 2020-09-17 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: HIV-1-infection; Gonorrhea Male; Chlamydia; Partner Communication
Keywords: Expedited Partner Therapy; MSM; Transgender women; HIV prevention; Peru
MeSH Terms: conditions — Chlamydia Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Expedited Partner Therapy (EPT) (Experimental): Participants in the EPT arm will receive up to five partner antibiotic treatment packets to deliver to their recent sexual partners following a diagnosis of gonorrhea (GC) and/or chlamydia (CT). The intervention will be repeated with all subsequent episodes of GC and/or CT infection during the 12-month follow-up period.
  Interventions: Behavioral: EPT
- Control (No Intervention): Participants in the control arm will receive standard-of-care counseling on partner notification following a diagnosis of gonorrhea (GC) and/or chlamydia (CT). The same counseling will be repeated with all subsequent episodes of GC and/or CT infection during the 12-month follow-up period.

INTERVENTIONS:
Behavioral: EPT — Expedited Partner Therapy (EPT) involves provision of empiric oral antibiotic therapy to the recent sexual partners of an individual diagnosed with gonorrhea and/or chlamydia infection.
  Arms: Expedited Partner Therapy (EPT)

SUMMARY:
The HIV epidemic in Peru remains concentrated in the subpopulation of men who have sex with men (MSM), where the prevalence of disease has been estimated between 10-22% in recent epidemiologic surveys. Partner-based methods to limit the spread of HIV and STI co-infection, including partner notification and partner treatment, provide an important new strategy for HIV control in the region.

Expedited Partner Therapy (EPT) has been shown to reduce rates of persistent or recurrent gonorrhea and chlamydia infection in heterosexual patients, but has not been fully evaluated for use among men who have sex with men (MSM). CDC guidelines support the use of EPT for partner management with heterosexual patients, but note the absence of evidence necessary to make an equivalent recommendation for the use of EPT with MSM. Randomized clinical trials to assess the impact of EPT on partner notification, treatment, and STI re-infection among MSM are critical to the development of evidence-based partner management guidelines.

As a theoretical model, EPT integrates behavioral, social, and biomedical approaches to HIV/STI control in a comprehensive prevention intervention. Our proposed exploration of the social and behavioral dimensions of partner notification and treatment will provide a methodological structure for understanding the influence of EPT on behavioral decision-making processes, interpersonal factors that influence partner notification, and network patterns of STI transmission within MSM populations in Peru.

The proposed study includes a screening protocol to identify eligible MSM subjects for participation in our planned study of the effect of EPT on partner notification, treatment, and linkage to HIV prevention and care services. Potential participants will complete a behavioral survey and undergo physical examination and testing for HIV, syphilis, gonorrhea, and chlamydia. Participants diagnosed with Gonorrhea and/or Chlamydia (at any anatomic site) will be eligible for enrollment in our Partner Management study of EPT and the HIV prevention cascade among MSM in Peru.

Participants in the Partner Management study will be randomly assigned to receive either standard of care partner notification counseling or standard counseling along with a maximum of five antibiotic treatment packets to deliver to their recent sexual partners. Participants will be asked to return to the site after 21 days to report on their actual partner notification behavior, with differences in notification evaluated between the two groups. Participants will then work with a study counselor to identify their recent partners and, if the participant agrees, to provide contact information so that the study team can contact these partners. Study staff will either confirm that the partner has already been notified, or provide notification of their likely STI exposure. After informing partners of their STI exposure, staff will ask partners to provide verbal consent to a single question evaluation (whether or not the partner had previously been informed of their exposure) to verify participant-reported behavior. Partners will also be asked to visit the study site to complete a brief survey of their sexual practices and treatment-seeking behavior, as well as to undergo testing for HIV and STIs. All of the above data will be used to construct models of the spread of HIV and STIs in local MSM networks, and the potential effect of EPT on controlling the spread of STIs in this population.

DETAILED DESCRIPTION:
Background and Objectives. Expedited Partner Therapy (EPT) provides a framework to integrate STI control with HIV prevention through the sexual networks of men who have sex with men (MSM). Partner notification, testing, and treatment are the critical first steps of an HIV prevention cascade that bridges partner notification with linkage to HIV prevention services and population-scale reductions in HIV/STI incidence. EPT has been shown effective in reducing risks for STI re-exposure among heterosexual men and women but remains controversial for use with MSM. Previous studies of EPT with heterosexual couples have demonstrated significant decreases in the risk of recurrence for gonorrhea (GC), chlamydia (CT) and other STIs. Objections to the use of EPT with MSM center on the prevalence of undiagnosed HIV and syphilis among their partners, and fears that providing access to antibiotics will discourage STI-exposed individuals from seeking additional treatment. However, the evidence-based foundation for these objections is limited. In our study of EPT for MSM with GC/CT in Peru, the odds of partner notification were significantly greater in the EPT arm (85.2%) than in the standard counseling arm (61.8%; OR=3.56). Additional research is needed to explore the use of EPT in MSM partnerships and to develop alternative conceptual frameworks capable of understanding the complex associations between EPT, STI control, and HIV prevention in MSM sexual networks. We hypothesize that EPT will increase the frequency of partner notification, encourage partners to seek HIV/STI counseling and testing, and promote linkage to HIV prevention and treatment services.

Differences in partnership formations and network structures of MSM necessitate correspondingly specific approaches to partner management. Heterosexual networks in previous partner therapy trials included a high frequency of stable or monogamous partnerships where HIV/STI risk could be localized and confined. In one study, the mean number of sexual partners in 3 months reported by men and women with GC/CT was 1.5. In another, 96% of women with CT named <2 recent partners, and most reported one. In these partnership contexts, EPT offers a simple method to control cyclical STI transmission in 2-core or 3-core networks of stable, recurrent sexual contacts. In contrast, sexual partnerships between MSM in the U.S. and Latin America are often part of large networks characterized by a diverse, concurrent mix of stable, casual, and anonymous partners. In a 2014 survey, MSM in Peru reported an average of 4.2 partners in the previous 30 days. The open structure of these decentralized, k-core networks limits the effectiveness of patient-delivered partner therapy in controlling cyclical STI re-transmission between stable partners. Instead, the primary benefit of EPT in these open-circuit networks lies in the potential to target HIV/STI prevention technologies to the highest risk nodes of diffuse and diverse sexual networks.

EPT offers an intervention ideally suited to Peru's local epidemiologic context. The Peruvian HIV epidemic is concentrated in the population of MSM and transgender women (TW) and associated with STI co-infection. In high-risk MSM populations, partner- and network-level characteristics have been found to be important factors contributing to HIV/STI acquisition. Sexual networks of at-risk MSM are often composed of a concurrent mix of stable/primary, casual (recurrent or single contact), anonymous, and/or commercial partners, with varying degrees of communication, trust, and responsibility. Although stable partners are considered "low-risk" for exposure to HIV/STIs, the lack of objective information on HIV/STI status and the increased likelihood of condomless intercourse in these partnership contexts lead to a high frequency of HIV/STI transmission. Casual sexual partners are often maintained concurrent with primary partners or anonymous contacts and contribute to the dissemination of HIV/STIs across diffuse social and geographic boundaries. Anonymous partners, by definition untraceable, are common and present significant challenges for STI control.

Previous research has emphasized how interpersonal contexts influence partner management tools. Internet systems encourage notification in casual partnerships with minimal interpersonal commitment and low perceived risk of re-exposure, while efforts to target prevention outreach to the dates and times of anonymous contacts have shown success. In contrast, EPT is most effective in stable or recurrent casual partnerships where trust and communication are assumed and the potential for STI re-exposure is high. While any comprehensive partner management strategy will require an array of systems to address the range of partnerships structuring MSM networks, EPT provides a critical tool to address HIV/STI transmission networks.

To evaluate the potential effectiveness of EPT for use with MSM, the investigators have identified three key questions:

i) What is the effect of EPT on self-reported behavioral notification practices and biological outcomes of recurrent GC/CT infection? ii) What is the effect of EPT on partner-confirmed notification outcomes, HIV/STI testing, and linkage to prevention/treatment services? and iii) Would observed increases in testing and treatment lead to reductions in population-level patterns of HIV/STI transmission?

Specific Aims Aim 1. To determine the effect of EPT on individual-level outcomes of partner notification and persistent or recurrent GC/CT infection among MSM. The investigators plan to recruit 2,208 behaviorally high-risk MSM from community-based HIV/STI testing sites to undergo nucleic acid testing for rectal, pharyngeal, and urethral GC/CT in order to identify 552 GC/CT-positive cases. Cases will be randomly assigned to receive standardized partner notification counseling, either alone or in combination with EPT (antibiotic treatment packets to deliver to their recent partners). Self-reported partner notification, associated factors including empowerment, stigma/ shame, barriers to partner testing/treatment, and prevalence of persistent or recurrent GC/CT will be compared between intervention and control arms at 21-Day Follow-up. To collect longitudinal data on post-intervention risk behavior and HIV/STI incidence, enrolled participants will be asked to return for quarterly HIV/STI testing over a 12-month period. Recurrent GC/CT cases will be managed according to the original randomization arm.

Aim 2. To assess the effect of EPT on partner-confirmed outcomes of notification, HIV/STI testing, STI treatment, and linkage to HIV prevention and treatment services. After completing the 21-Day Follow-up evaluation, participants will be asked to provide partner contact information for study staff to confirm participant-reported outcomes. Assessments will be conducted by telephone, and partners will be asked to visit the site for HIV, syphilis, and GC/CT testing and to complete a brief survey of their post-notification behavior, including subsequent HIV/STI testing, STI treatment, and uptake of HIV prevention and treatment services.

Aim 3. To model the impact of EPT for partners of MSM on network- and community-level patterns of HIV and STI transmission. Empiric data from Aims 1 and 2, supplemented by data from published literature, will be used to construct Agent-Based Models estimating the effect of observed individual- and partner-level outcomes on projected population-level HIV/STI transmission. Empiric data on the effect of EPT on prevention cascade outcomes of partner notification, HIV/STI testing, antibiotic treatment, and uptake of biomedical prevention methods like PrEP and TasP, and subsequent observations of GC/CT prevalence and incidence, as well as cohort patterns of HIV and STI acquisition, re-infection, and co-transmission will all be collected. These data points will be used to inform population-scale models comparing HIV incidence in the intervention and control arms and to assess the community-level impact of EPT on STI control and HIV prevention.

Study Design and Methods Overview. The investigators will conduct a randomized controlled trial to assess the effect of Expedited Partner Therapy (EPT) on self-reported partner notification and recurrent GC/CT infection among MSM with GC/CT (Figure 1).

Based on prior studies among MSM in Peru where GC/CT prevalence was 30-40%, the investigators anticipate screening 2,208 men to recruit a cohort of 552 GC/CT-infected MSM [101, 128, 129]. Screening procedures will include assessment of demographic and behavioral characteristics, and HIV, syphilis, and GC/CT testing.

I. Screening. Screening procedures will assess for eligibility and obtain baseline HIV/STI prevalence data for the population. In order to assess for HIV acquisition and transmission risk, and to map mixing patterns by HIV status within sexual networks, both HIV-infected and -uninfected MSM will be eligible. Due to significant differences in partnership structures, interactions, and notification practices between MSM and transgender women (TW), only MSM will be enrolled. Screening will continue until enrolling 552 GC/CT-infected MSM.

i) Behavioral Survey: All screened participants will be asked to complete an ACASI survey assessing demographics, substance use, history of HIV/STI testing, use of PrEP (if HIV-uninfected) or antiretroviral therapy (if HIV-infected), sexual practices, characteristics of recent partners, and sexual network composition.

ii) Rapid HIV Testing: Study staff will provide pre- and post-test HIV risk reduction counseling based on the CDC's RESPECT-2 model and screen for HIV with a 4th Generation Rapid HIV-1/2 assay (Alere Determine, Alere) [130]. Participants with a positive rapid test will be informed of their results and a blood sample will be sent for confirmatory Western Blot testing. Referrals to HIV prevention and treatment services (including PrEP and ART) offered at Via Libre and other local sites will be provided according to the participant's serostatus.

iii) Viral Load Testing. In order to assess the burden of HIV viremia (and risks for secondary HIV transmission) in the population, samples for HIV-1 PCR testing will be collected from all HIV-infected participants at Screening.

iv) Physical Examination: Participants will undergo routine physical examination to assess for signs of untreated STIs. Participants with primary or secondary syphilis or with a known exposure to syphilis, will be treated with Benzathine Penicillin G 2.4 million IU (or, if allergic to Penicillin, with Doxycycline 100 mg PO BID x 7 days). Participants with urethral and/or rectal discharge or inflammation will be treated with Ceftriaxone 250 mg IM and Doxycycline 100 mg PO BID x 7 days.

v) Syphilis Testing: Participants will undergo syphilis testing by RPR (RPRnosticon, Biomerieux), with positive results confirmed by TPPA (Serodia TPPA, Fujirebio) and serial dilution of positive titers. Individuals with latent syphilis diagnosed by laboratory testing will be treated with three weekly IM doses of Penicillin G or a 21 day course of oral Doxycycline (100 mg PO BID), if allergic to Penicillin.

vi) GC/CT Nucleic Acid Testing: All participants will be tested for pharyngeal, rectal, and urethral GC/CT. First-catch urine samples will be self-collected by participants. Pharyngeal and rectal swabs will be obtained by clinical staff. (Participants will also be allowed to self collect rectal swab samples, if preferred.) Samples will be tested for GC/CT using a transcription mediated assay (TMA) (GenProbe Aptima, Hologic). Results of laboratory testing will be provided within 14 days at a scheduled Follow-up visit. Participants with asymptomatic GC/CT will be provided with appropriate antibiotic treatment (Ceftriaxone 250 mg IM and Doxycycline 100 mg PO BID x 7 days for GC or GC/CT co-infection; Doxycycline 100 mg PO BID x 7 days for CT mono-infection). While no specific follow-up testing will be performed, all participants will be encouraged to seek routine STI screening in 3-6 months, according to their sexual risk behavior. Study protocols for antibiotic treatment and follow-up testing are consistent with the US CDC 2015 Recommendations for STI Treatment.

vii) Follow-up Visit: All participants will be asked to return for a Follow-up visit within 14 days to receive results of laboratory testing.

viii) Enrollment: Participants with symptomatic urethritis/proctitis at the Initial Visit or with laboratory diagnosed GC/CT infection (at any anatomic site) at the Follow-up visit will be eligible for randomization.

vii) Randomization: Eligible participants will be randomly assigned to intervention and control arms on a 1-to-1 basis. Assignments will be generated through the site www.random.org in random permuted blocks of 5. Assignments will be stored in sealed envelopes to be opened and recorded at enrollment.

viii) Anticipated Partner Notification Survey: After randomization, participants will be asked to complete a survey assessing partner notification attitudes, beliefs, and anticipated practices. The survey instrument has been developed from our previous work with MSM in Peru and addresses behavioral, biological, and social factors associated with notification.

1. Behavioral Factors: Introductory questions address behavioral, normative, and control beliefs associated with PN and are based on previous qualitative research with MSM in Peru. Previously developed and validated scales addressing STI stigma and shame, partner notification and condom use self-efficacy, depression, anxiety, and substance use will provide information on behavioral contexts of notification decisions. A Spanish version of the Marlowe-Crowne Social Desirability Scale will be used to assess for response bias.
2. Biomedical Factors: Biological characteristics of the individual, the pathogen, and the partnership will be used to evaluate for presence or absence of symptoms, perceived risks of having infected (or been infected by) a given partner, and risk of secondary HIV/STI transmission.
3. Social Factors: Sexual network characteristics, including the gender and sexual identity of the participant and their recent partner(s), partnership type, and partner-specific risk behavior will be assessed. Survey questions ask about participants' sexual behavior (including condomless insertive and receptive anal intercourse with serodiscordant or unknown status partners), and substance use. To assess partner-specific factors, participants will be asked to described characteristics of their three most recent sexual contacts, sexual practices with these partners, anticipated likelihood of notifying each partner, and incentives or barriers to notification. In order to assist with future recall, participants will be asked to provide a name, nickname, or identifying characteristic (e.g., "The guy in the blue shirt from Vale Todo") for each of these partners.

ix) Partner Notification Counseling: All participants will be provided with partner notification counseling using a standardized script. The scripted message will advise the recipient of the importance of informing recent sexual partners of their diagnosis, and the availability of free partner testing at the Via Libre site.

x) Expedited Partner Therapy: Participants assigned to the EPT arm will also be provided with a maximum of 5 EPT partner treatment packets. The number of packets is limited in order to reduce the risk of diversion or inappropriate use of antibiotics while still providing reasonable partner access to treatment. Each packet will contain single doses of Cefixime (400 mg) and Azithromycin (1g), as well as Spanish-language printed information on GC/CT infection and local sites offering free or low-cost HIV/STI testing and treatment (including Via Libre). (Cefixime is recommended by the CDC as an oral treatment option for GC infection in situations where use of injectable ceftriaxone is not feasible, for instance in cases of partner-delivered antibiotic therapy.) Printed information will include a message advising the recipient that they are at high risk of exposure to HIV, syphilis, and GC/CT, that they should seek HIV/STI testing and treatment at a local health care facility, and that they should only take the antibiotics provided if they are unable or unwilling to seek appropriate care. Participants will be counseled by study staff on the proper use and distribution of partner treatment packets using a pre-scripted message.

xi) 21-Day Follow-Up Assessment: 21 days after diagnosis, participants with GC/CT infection will be asked to return to the clinic for a Follow-up Visit including survey assessment of partner notification and treatment outcomes and biological test of cure.

Behavioral Outcomes Survey. Participants will be asked to complete an ACASI Partner Notification Outcomes survey. Participants will be reminded of the number of recent sexual partners they reported on the Enrollment Survey and asked to describe both how many of these partners were notified of their GC/CT diagnosis and how many partners were provided with EPT treatment packets (if applicable). Participants will be reminded of the basic characteristics of their 3 most recent sexual partners (gender, sexual identity, and first name or other label used to identify the partner) and asked to state whether each of these partners was notified, whether they received antibiotic therapy (either from the participant or from a different source), whether they received testing for HIV and other STIs, and why each partner was or was not informed of their STI exposure.

Biological Test of Cure. Repeat TMA testing for GC/CT infection will be conducted only at the site of the initial GC/CT infection, with results provided by phone or in person within 14 days. Participants with persistent or recurrent infection will be provided with an additional course of antibiotic therapy. Confirmation of Notification. After completing Follow-up assessments, counselors will interview participants to review partner notification outcomes and to request partner contact information to confirm reported outcomes. Procedures for participant interviewing and partner contact are described below (Aim 2).

II. Quarterly Monitoring Visits. i. Monitoring Procedures. Participants will be asked to return to the study site every three months (starting from the date of their initial Screening Visit) over a 12-month period for repeat HIV/STI testing and re-assessment of sexual behavior and network patterns. Participants will be asked to complete a brief, ACASI-administered survey at each visit. Similar to the Baseline survey, the Monitoring questionnaire will assess sexual risk behavior, substance use, sexual partnerships, and sexual network characteristics during the previous 3-month interval. Participants will also undergo physical examination for signs or symptoms of STIs following the procedures outlined above. Rapid HIV and syphilis testing will be performed at each visit using the procedures outlined above. Repeat testing for pharyngeal, rectal, and urethral GC/CT infection will be performed at each visit with results provided by telephone or in person within 14 days.

ii. Repeat Episodes of GC/CT. Recurrent cases of GC/CT infection will be managed according to the procedures listed above. Participants diagnosed with recurrent GC/CT will be asked to come to the clinic site for treatment with Ceftriaxone 250 mg IM and/or Doxycycline 100 mg PO BID for 7 days. Partner management procedures will be delivered according to the original randomization assignment. Participants in the Control arm will receive standardized Partner Notification counseling as described above. Participants assigned to the EPT arm will be provided with an additional set of 5 partner treatment packets. Participants in both arms will be asked to complete the Anticipated Partner Notification Survey as described above.

iii. Follow-Up Assessment: Participants with recurrent GC/CT will be asked to return for additional 21-Day Follow-Up Assessment(s). At the Follow-up visit, participants will be asked to complete the Partner Notification Outcomes survey, to undergo test of cure for GC/CT, and to provide partner contact information.

III. Aim 2 will focus on partner confirmation of notification and treatment outcomes, and biological assessment of partner HIV/STI status. After completing 21-Day Follow-up procedures, participants will be asked for permission to contact their recent sexual partners in order for study staff to confirm reported notification outcomes (or to advise uninformed partners of their exposure). Counselors will attempt to contact recent partners by telephone, inform them of their STI exposure, and ask them to visit the study site for a single visit including HIV/STI testing, completion of a behavioral survey, and appropriate antibiotic treatment.

i. Contact Tracing. After completing the 21-Day Follow-up assessment, participants with GC/CT will undergo a partner notification interview with study staff. Counseling sessions will draw on established practices for partner recall in STI interviewing, in accordance with Peruvian Ministry of Health guidelines. Assessments will use Timeline Follow-Back (TLFB) methods to generate a detailed accounting of all sexual partners during the 60-day period prior to diagnosis. Counselors will work with participants to enumerate their total number of sexual partners, identify all named partners, and elicit available contact information. Although participants will be advised that notification will be conducted anonymously, without revealing their name or other identifying characteristics, the possibility of partner violence or other negative responses to notification will be discussed. Participants will be given the option to decline to provide contact information for any partner(s) they do not wish to inform.

ii. Partner Notification and Telephone Survey. Counselors will attempt to contact named partners by telephone to inform them of their exposure to GC/CT, to discuss the importance of HIV/STI testing, and to advise them of the availability of free testing at the study site. After answering any questions, counselors will ask for consent to conduct a brief telephone survey. If agreed, the counselor will administer a 5-question survey of whether the partner had been notified of their STI exposure, how they were notified and/or who notified them), if they received antibiotic treatment, how they received the treatment, and whether they sought HIV/STI testing. Partners will be invited to the study site for HIV/STI testing and additional study procedures.

iii. Partner Clinic Assessment. Partners who visit the study site will participate in a single-session evaluation of notification and treatment outcomes. Partners will be asked to complete an ACASI survey describing their demographic information, sexual behavior, HIV/STI history, number and type of all recent sexual partners, and characteristics of their three most recent sexual partners. After completing the survey, partners will be examined for signs or STIs and tested for HIV, syphilis, and GC/CT using the procedures described above. Viral load testing will be performed for partners with new or previously diagnosed HIV infection. Results of laboratory testing will be provided within 14 days. Appropriate antibiotic treatment and/or referrals for HIV prevention and treatment services will be provided to all partners based on HIV/STI status as described above.

ELIGIBILITY:
Inclusion Criteria:

1. Anatomically male at birth
2. Condomless anal intercourse with an HIV serodiscordant or unknown serostatus male or transgender female partner in the previous 6 months
3. 18 years of age or older
4. Diagnosis of Gonorrhea and/or Chlamydia infection at any anatomic site at the Screening visit

Exclusion Criteria:

1) Inability to understand the study procedures or to provide informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 555 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Self-reported partner notification | 21 Days
  Participant self-report of notification of one or more sexual partners at 21-days Follow-up
Partner-confirmed notification | 60 Days
  Confirmation by named partners following notification of STI exposure by the index participant

SECONDARY OUTCOMES:
Self-reported partner treatment | 21 Days
  Participant self-report of antibiotic treatment of one or more sexual partners at 21-days
Self-reported partner HIV/STI testing | 21 Days
  Participant self-report of HIV/STI testing by one or more sexual partners at 21-days
Partner confirmed treatment | 60 Days
  Partner confirmation of antibiotic treatment following notification of STI exposure by the index participant
Partner confirmed HIV/STI testing | 60 Days
  Partner confirmation of HIV/STI testing following notification of STI exposure by the index participant

CONTACTS AND LOCATIONS:
Overall Officials: Jesse L Clark, MD, MSc, Principal Investigator — Associate Professor-in-Residence
Locations (1):
- Asociacion Civil Via Libre, Lima, Peru

IPD SHARING:
Plan to Share IPD: No